





# Exercise Snacking to Improve Strength and STability: ESISST pilot study

#### **Informed Consent Form**

### Investigators

Dr Oly Perkin

Dr Max Western

Dr Tomas Welsh

(O.J.Perkin@bath.ac.uk)

(M.J.Western@bath.ac.uk)

(tw695@bath.ac.uk)

| | | initial box |
|---|---|---|
| 1. | I confirm that I have read the participant information sheet and I have had the opportunity to consider the information, ask questions, and have satisfactory answers. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | |
| 3. | I understand that I will be asked to undertake two bouts of homebased exercise snacking a day for 28 consecutive days | |
| 4. | I understand who will have access to the data, how the data will be stored, what will happen to the data at the end of the project, and that if I wish to withdraw my data from the project I must inform the investigators before publication of the findings. | |
| 5. | I understand that this project has received ethical approval from the NHS South West – Frenchay Research Ethics Committee [reference: 22/SW/0084]. | |
| 6. | I agree that a copy of this informed consent form will be stored at<br>the Research Institute for Care of Older People for 10 years in<br>accordance with the University of Bath's Data Retention Policy as<br>Sponsor of the research. | |

| [ | Date: | <u>Partici</u> | oant Copy |
|---|---|---|---|
| F | Researcher Signature: | | |
| F | Researcher Name: | | |
| | Date: | | |
| F | Participant Signature: | | |
| F | Participant Name: | | |
| iii) | I agree to take part in the optional audio-recorded interview at the end of the study, but I understand that I can change my mind nearer the time. | | |
| ii) | I give permission for my GP to be informed that I am participating in this study (this is optional). | | |
| i) | I give permission to the University of Bath Research<br>Data Archive to grant access to this anonymous data<br>to support ethically approved research in the future. | | |
| <u>Opti</u> | onal questions | Yes | No |
| 8. | I agree to take part in the above study. | | |
| 7. | 7. I agree that the anonymous data collected in this study, will be stored in the University of Bath Research Data Archive for 10 years from the point that data collection is complete, after which point it will be destroyed in accordance with the University of Bath's Data Retention Policy. | | |







# Exercise Snacking to Improve Strength and STability: ESISST pilot study

#### **Informed Consent Form**

#### **Investigators**

Dr Oly Perkin

Dr Max Western

Dr Tomas Welsh

(O.J.Perkin@bath.ac.uk)

(M.J.Western@bath.ac.uk)

(tw695@bath.ac.uk)

| | | initial box |
|---|---|---|
| 1. | I confirm that I have read the participant information sheet and I have had the opportunity to consider the information, ask questions, and have satisfactory answers. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | |
| 3. | I understand that I will be asked to undertake two bouts of homebased exercise snacking a day for 28 consecutive days | |
| 4. | I understand who will have access to the data, how the data will be stored, what will happen to the data at the end of the project, and that if I wish to withdraw my data from the project I must inform the investigators before publication of the findings. | |
| 5. | I understand that this project has received ethical approval from the NHS South West – Frenchay Research Ethics Committee [reference: 22/SW/0084]. | |
| 6. | I agree that a copy of this informed consent form will be stored at<br>the Research Institute for Care of Older People for 10 years in<br>accordance with the University of Bath's Data Retention Policy<br>as Sponsor of the research | |

| D | ate: | Site File | e Copy |
|---|---|---|---|
| R | esearcher Signature: | | |
| R | esearcher Name: | | |
| D | ate: | | |
| Pa | articipant Signature: | | |
| Pa | articipant Name: | | |
| iii) | I agree to take part in the optional audio-recorded interview at the end of the study, but I understand that I can change my mind nearer the time. | | |
| ii) | I give permission for my GP to be informed that I am participating in this study (this is optional). | | |
| i) | I give permission to the University of Bath Research Data Archive to grant access to this anonymous data to support ethically approved research in the future. | | |
| <u>Optio</u> | nal questions | Yes | No |
| 8. | I agree to take part in the above study. | | |
| 7. | 7. I agree that the anonymous data collected in this study, will be stored in the University of Bath Research Data Archive for 10 years from the point that data collection is complete, after which point it will be destroyed in accordance with the University of Bath's Data Retention Policy. | | |







### Exercise Snacking to Improve Strength and STability: ESISST pilot study

#### **Informed Consent Form**

### Investigators

Dr Oly Perkin

Dr Max Western

Dr Tomas Welsh

(O.J.Perkin@bath.ac.uk)

(M.J.Western@bath.ac.uk)

(tw695@bath.ac.uk)

| | | Please initial box |
|---|---|---|
| 1. | I confirm that I have read the participant information sheet and I have had the opportunity to consider the information, ask questions, and have satisfactory answers. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | |
| 3. | I understand that I will be asked to undertake two bouts of homebased exercise snacking a day for 28 consecutive days | |
| 4. | I understand who will have access to the data, how the data will be stored, what will happen to the data at the end of the project, and that if I wish to withdraw my data from the project I must inform the investigators before publication of the findings. | |
| 5. | I understand that this project has received ethical approval from the NHS South West – Frenchay Research Ethics Committee [reference: 22/SW/0084]. | |
| 6. | I agree that a copy of this informed consent form will be stored at<br>the Research Institute for Care of Older People for 10 years in<br>accordance with the University of Bath's Data Retention Policy<br>as Sponsor of the research | |

| | Da | te: | Medical R | ecords Copy |
|---|---|---|---|---|
| | Re | searcher Signature: | | |
| | Re | searcher Name: | | |
| | Da | te: | | |
| | Pa | rticipant Signature: | | |
| | Pa | rticipant Name: | | |
| | iii) | I agree to take part in the optional audio-recorded interview at the end of the study, but I understand that I can change my mind nearer the time. | | |
| | ii) | I give permission for my GP to be informed that I am participating in this study (this is optional). | | |
| | i) I | give permission to the University of Bath Research<br>Data Archive to grant access to this anonymous<br>data to support ethically approved research in the<br>future. | | |
| <u>C</u> | otior | nal questions | Yes | No |
| | 8. | I agree to take part in the above study. | | |
| | 7. | I agree that the anonymous data collected in this s<br>stored in the University of Bath Research Data A<br>years from the point that data collection is complete<br>point it will be destroyed in accordance with the<br>Bath's Data Retention Policy. | rchive for 1<br>e, after whic | o<br>ch |